CLINICAL TRIAL: NCT03242538
Title: Prehabilitation for Port Films: Phase 1. Evaluating Orthopedic Measurements of Pelvic Tilt During Radiation Treatments for Pelvic Cancer
Brief Title: Prehabilitation for Pelvic Cancer: Changes in Setup Variability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Responsible Party: Principal Investigator, Janaki Moni, Associate Professor, Department of Radiation Oncology, University of Massachusetts, Worcester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: H00013328
Record Dates: First submitted 2017-07-31; First posted 2017-08-08 (Actual); Last update posted 2019-09-11 (Actual); Status verified 2019-09

CONDITIONS: Pelvic Cancer
Keywords: Exercise
MeSH Terms: conditions — Pelvic Neoplasms; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pelvic Exercise Intervention (Experimental): Patients will perform two pelvic exercises prior to each external beam radiation treatment.
  Interventions: Behavioral: Pelvic Exercise

INTERVENTIONS:
Behavioral: Pelvic Exercise — Hip extension and external hip rotation exercises are completed prior to daily external beam radiation treatment.

SUMMARY:
The investigators hypothesize that two pelvic relaxation exercises will be feasible and safe to perform by subjects daily before radiation during the participant's treatment and will decrease variability of sacral slope measurements on daily port films. The investigators will observe trends in the daily variability and change in the sacral slope in each participant to determine if this could decrease variability. The investigators will compare these measurements to a retrospective cohort that did not have the exercises, but did demonstrate variability. Reducing set-up variability (which inadvertently occurs during radiation) is important to improve radiation targets and diminish potential adverse effects. The investigators will query participants for objective and subjective feedback on the exercises and record frequency and duration of the two exercises.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be >21 yrs of age and will have an oncologic diagnosis that requires a course of pelvic radiation therapy for a minimum of 5 weeks.
* They will have an ECOG Performance Status (This scale, developed by the Eastern Cooperative Oncology Group (ECOG), now part of the ECOG-ACRIN (American College of Radiology Imaging Network) Cancer Research Group, describes a patient's level of functioning in terms of their ability to care for themselves, daily activity, and physical ability (walking, working, etc.)) of 1 or better as determined by patient history.
* They will be ambulatory without needing any ambulatory aids such as a cane or walker.
* Both men and women will be eligible as there is no significant anatomical difference in sacral slope measurement. Joint replacement patients will not be excluded.

Exclusion Criteria:

* Adults unable to consent
* Individuals who are not yet adults (infants, children, teenagers)
* Pregnant women
* Prisoners
* Non-English speaking subjects

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2017-06-23 (Actual); Primary Completion 2018-07-21 (Actual); Study Completion 2019-01-17 (Actual)

PRIMARY OUTCOMES:
Sacral Slope Variation | Daily, through duration of radiation treatment, averaging 6-10 weeks
  Reduced variation in sacral slope angle measured on daily port films.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Baima, MD, Principal Investigator — UMass Medical - Department of Orthopedics; Janaki Moni, MD, Principal Investigator — UMass Medical - Department of Radiation Oncology
Locations (1):
- University of Massachusetts Medical School, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] O'Loughlin L, Lukez A, Ma Y, Baima J, Moni J. Prehabilitation for patient positioning: pelvic exercises assist in minimizing inter-fraction sacral slope variability during radiation therapy. Med Oncol. 2019 Nov 12;37(1):3. doi: 10.1007/s12032-019-1322-9. PMID 31713056